CLINICAL TRIAL: NCT06404619
Title: Impact of mHealth Implementation Program on Improving Nursing Students' Lifestyle: A Randomized Controlled Trial
Brief Title: Impact of mHealth Implementation Program on Improving Nursing Students' Lifestyle
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Shaherah Andargeery, Principal Investigator, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PNURSP2024R447
Record Dates: First submitted 2024-04-23; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy Lifestyle
Keywords: lifestyle; mHealth; nursing student
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth education program (Experimental): They received 1 session every 2 weeks for 3 months using Zoom meeting (each session lasts for 1 hour). The message emphasizes the importance of quality of life and positive psychology and highlights the steps to change one's lifestyle, including self-reflection, habit modification, and commitment to a comprehensive lifestyle change include importance of physical activity, management of stress, quality and quantity of sleep and specific recommendations are provided regarding drinking water, organizing meals, and adopting a healthy balanced diet with attention to portion sizes. Daily engagement with the intervention was assessed using text message replies and number of coaching calls completed. Participants were asked to reply "Done" via Emails, Facebook, WhatsApp, Telegram, Instagram, or Zoom meeting.
  Interventions: Behavioral: Education program
- Traditional education program (Active Comparator): They received 1 session every 2 weeks for 3 months at their convenience place (each session lasts for 1 hour). The same message as the Intervention group. Small group discussions and display of educational messages, posters, handout, and power point presentation lectures.
  Interventions: Behavioral: Education program

INTERVENTIONS:
Behavioral: Education program — The message emphasizes the importance of quality of life and positive psychology. The concept of quality of life is described as multidimensional, also the message highlights the steps to change one's lifestyle, including self-reflection, habit modification, and commitment to a comprehensive lifestyle change include importance of physical activity, management of stress, quality and quantity of sleep and specific recommendations are provided regarding drinking water, organizing meals, and adopting a healthy balanced diet with attention to portion sizes. The message also discussed fitness foods that aid digestion and promote a healthy body. The message introduced the Healthy Eating Plate.

SUMMARY:
Healthy lifestyles are crucial for preventing chronic diseases. This study evaluated the effectiveness of mHealth intervention program in adopting healthy lifestyles.

DETAILED DESCRIPTION:
Healthy lifestyles are crucial for preventing chronic diseases. Nonetheless, approximately 90% of university students regularly engage in at least one unhealthy lifestyle. Mobile smart devices-based health interventions (mHealth) that incorporate theoretical frameworks regarding behavioral change in interaction with the environment may provide an appealing and cost-effective approach for promoting sustainable adaptations of healthier lifestyles.

The aim of this study was to evaluate the effectiveness of mHealth intervention program compared to traditional (face-to-face) program in adopting healthy lifestyles among students of the Faculty of Nursing.

ELIGIBILITY:
Inclusion Criteria:

* male or female nurse student
* aged 19-24 years
* with BMI ≥ 18.5
* capable of performing physical activity
* owner of a smartphone
* ready to use different social media

Exclusion Criteria:

* on diet regimen or have a history of diet regimen
* with history of chronic diseases e.g., DM, hypothyroidism or other endocrinal diseases
* with history of medications that may cause weight gain e.g., antipsychotics, antidepressants, antiepileptics or steroids
* with mental or psychological disorders

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity time and levels of participants as assessed by Global/International Physical Activity Questionnaire (GPAQ/IPAQ). | Assessed just before and immediately after the intervention
  The total weekly time spent on physical activity and the time spent in each domain (work, transportation, and recreational time) are determined by multiplying the number of days per week in each category by the average daily duration. Minutes per week in each category are then multiplied by metabolic equivalents (MET). The overall GPAQ score is described as "Low" if < 600 MET-minutes/week, "Moderate" if = 600-1500 MET-minutes/week, or "High" if > 1500 MET-minutes/week.
Dietary assessment using Food frequency questionnaire (FFQ). | Assessed just before and immediately after the intervention
  It consists of 140 food items categorized under 27 categories with three Likert scale (usually eat, sometimes eat, and rarely eat). Score of 27-45 indicates bad healthy choices, 46-63 indicate fair healthy choices, and 64-81 indicate good healthy choices.
Sleep quality scale. | Assessed just before and immediately after the intervention
  It assesses the quality of sleep for the last one month and consists of 28 questions with four Likert scale (rarely, sometimes, often, and almost always). The total score can range from 0 to 84, with higher scores demoting more more frequent sleep disturbances (Good quality of sleep ≤ 28, Fair 29 - ≤ 56, and poor > 56).

SECONDARY OUTCOMES:
The weight in kilograms and height in meters will be combined to report the body mass index (BMI) in kg/m2. | Assessed just before and immediately after the intervention
  Participants are categorized according to the BMI according to WHO into:
  * Underweight (BMI < 18.5 kg/m2)
  * Normal weight (BMI = 18.5 - 24.9 kg/m2)
  * Overweight (BMI = 25 - 29.9 kg/m2)
  * Obese (BMI ≥ 30 kg/m2)
Blood Pressure Level assessed with the sphygmomanometer. | Assessed just before and immediately after the intervention
  Participants are categorized according to their blood pressure into:
  * Normal blood pressure: Less than 120/80 mmHg
  * At risk for high blood pressure (prehypertension): Between 120/80 and 140/90
  * High blood pressure (hypertension): More than 140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Shaherah Andargeery, MD, Principal Investigator — College of Nursing, Princess Nourah bint Abdulrahman University
Locations (1):
- College of Nursing Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
We will share the individual de-identified participants' data. The datasets generated during and/or analyzed during the current study will be available from the corresponding author on reasonable request, beginning 12 months and ending 36 months following article publication.
Supporting Information: Study Protocol
Time Frame: Between 12 and 36 months after article publication
Access Criteria: Data will be accessible to researchers to be used for systematic reviews or meta-analyses based on a reasonable request to the corresponding author.

REFERENCES:
- [Derived] Andargeery SY, El-Rafey DS. A randomized controlled trial of the effectiveness of the mHealth program in improving the lifestyle of nursing students. Sci Rep. 2025 Mar 21;15(1):9765. doi: 10.1038/s41598-024-80982-2. PMID 40118869